CLINICAL TRIAL: NCT06733363
Title: A Scalable Cruciferous Vegetable Intervention to Reduce Bladder Cancer Recurrence and Progression
Brief Title: A Cruciferous Vegetable Eating Program for the Reduction of Cancer Recurrence and Progression in Patients With Non-muscle Invasive Bladder Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: I-4207024; R01CA296175 (NIH)
Record Dates: First submitted 2024-12-10; First posted 2024-12-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Non-Muscle Invasive Bladder Carcinoma; Recurrent Bladder Carcinoma; Recurrent Non-Muscle Invasive Bladder Carcinoma; Stage 0a Bladder Cancer AJCC v8; Stage 1 Bladder Cancer AJCC v8
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms; Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The Data Collector will be masked to treatment assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adaptation (Experimental): CAB members participate in maintenance phase development discussion over an hour up to 3 times per week.
  Interventions: Behavioral: Behavioral Dietary Intervention
- Arm II - POW-R Health Only/Core + Maintenance (Experimental): Patients receive study materials and phone calls during life of study
  Interventions: Behavioral: Telephone- Based Intervention

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Participate in POW-R Health Only/Core program
  Arms: Adaptation
Behavioral: Telephone- Based Intervention — Receive live phone calls
  Arms: Arm II - POW-R Health Only/Core + Maintenance

SUMMARY:
This phase II trial is being done to develop and test a healthy eating program to reduce cancer recurrence (cancer that has come back after a period of improvement) and/or progression (cancer that is growing, spreading, or getting worse) in patients with non-muscle invasive bladder cancer (NMIBC). Researchers want to better understand how incorporating more cruciferous vegetables in the diet may reduce the risk of cancer recurrence or progression in men and women who were diagnosed with early-stage bladder cancer and compare whether extending the program can further improve bladder cancer outcomes. POW-R Health is a behavioral dietary intervention designed to modestly increase cruciferous vegetable (cruciferae) intake in patients. Cruciferous vegetables, such as cabbage, kale and broccoli, arugula, contain phytochemicals known as isothiocyanates (ITCs). Dietary ITCs exert potent anticancer activities against bladder cancer and can be rapidly metabolized, delivered to the bladder, and concentrated in the urine. Participating in the healthy eating program may reduce bladder cancer recurrence or progression in NMIBC survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop a maintenance component to add onto our POW-R Health intervention (POW-R Health Only/Core) to create POW-R Health + Maintenance.

II. Assess the efficacy of POW-R Health + Maintenance compared to POW-R Health Only/Core using a 2-group randomized controlled trial (RCT) design in 344 participants on the primary outcome of urinary ITC.

SECONDARY OBJECTIVE:

I. Assess the efficacy of POW-R Health + Maintenance compared to POW-R Health Only/Core on the secondary outcome of cruciferae intake.

ELIGIBILITY:
Inclusion Criteria:

* English speaking

  * Diagnosed with stage Tis, Ta, or T1 bladder cancer
  * Age 18 years old or older (no upper limit)
  * Resides in New York State
  * Cancer not reported by a lab, nursing home, or death certificate/autopsy only
  * Did not receive a partial or radical cystectomy
  * Does not have other cancer diagnosis within 12 month of bladder cancer diagnosis nor under active treatment for any other cancers

Exclusion Criteria:

* Participants who had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

  * Adults unable to consent
  * Adults unable to complete study measures in English
  * Individuals who are not yet adults (infants, children, teenagers)
  * Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
  * Unwilling or unable to follow protocol requirements
  * The following special populations ae excluded from this study:

    * Cognitively impaired adults/adults with impaired decision-making capacity
    * Individuals who are not yet adults (infants, children, teenagers)
    * Pregnant women
    * Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 344 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2028-01-13 (Estimated); Study Completion 2029-02-28 (Estimated)

PRIMARY OUTCOMES:
Urinary isothiocyanates (ITCs) levels | Baseline throughout life of study - up to 24 months
  Levels with be measured using high performance liquid chromatography-based cyclocondensation assay

SECONDARY OUTCOMES:
Increase in Cruciferae Intake | up to 24 months
  Increase in Cruciferae Intake

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeary, MD, Principal Investigator — Roswell Park Comprehensive Cancer Center
Locations (1):
- Roswell Park Comprehensive Cancer Center, Buffalo, New York, United States